CLINICAL TRIAL: NCT01332383
Title: Special Drug Use Investigation for AMERGE Tablet (Long-term)
Brief Title: Special Drug Use Investigation for AMERGE® Tablet (Long-term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112925
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — naratriptan

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed AMERGE: Patients with migraine disorders prescribed AMERGE during study period
  Interventions: Drug: Naratriptan

INTERVENTIONS:
Drug: Naratriptan

SUMMARY:
To investigate the long-term safety and efficacy of AMERGE (naratriptan hydrochloride) on Japanese patients with migraine headache in clinical setting

ELIGIBILITY:
Inclusion Criteria:

* Must use AMERGE for the first time

Exclusion Criteria:

* Patients with hypersensitivity to naratriptan or any of the components.
* Patients with history, symptoms, or signs of myocardial infarction, ischemic cardiac or angina inversa
* Patients with history of cerebral vascular disturbance or transient ischaemic attack
* Patients with peripheral vascular syndromes
* Patients with uncontrolled hypertension
* Patients with severe renal or hepatic impairment
* Patients using treatment with another 5-HT1 agonist, an ergotamine-containing or ergot-type medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with migraine headache who are naive to AMERGE
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of adverse drug reactions and serious adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline